CLINICAL TRIAL: NCT03928444
Title: Evaluation of the Efficacy and Tolerability of Autologous Adipose Tissue Derived Stem Cells on Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Aliaa Ismail Ali Ismail, principle investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlexandriaUdermatology
Record Dates: First submitted 2019-04-21; First posted 2019-04-26 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Skin Rejuvenation
Keywords: Adipose tissue derived stem cells; Facial rejuvenation

STUDY DESIGN:
Intervention Model Description: split face
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stem cells (Experimental): one side of the face to be treated with intradermal stem cells
  Interventions: Procedure: intradermal injection of adipose derived stem cells to one side of the face
- control (Placebo Comparator): one side of face treated with intradermal saline
  Interventions: Procedure: intradermal injection of saline to one side of the face

INTERVENTIONS:
Procedure: intradermal injection of adipose derived stem cells to one side of the face — Lipoaspiration for preparation of ADSC will be done according to the following technique:
  Under local anesthesia using strict aseptic technique, a small incision will be done in the lateral aspect of the thigh or lower abdomen, through which the infiltration cannula will be introduced to inject the local anesthetic solution using the wet technique. This will be followed 15 minutes later by lipo-aspiration of (50 ml fat ) using a blunt tipped cannula under the negative suction pressure of a 60 ml syringe.
  * Autologous adipose tissue derived stem cells (At-ADSCs) will be separated from the lipo-aspirate using enzymatic digestion and differential centrifugation in the Center of Excellence for Research in Regenerative Medicine and its Application (CERRMA), Alexandria Faculty of Medicine.
  * Viability of collected cells will be checked using trypan blue stain. Characterization of the isolated ADSCs population will be performed by flow cytometry.
  Arms: stem cells
Procedure: intradermal injection of saline to one side of the face — intradermal injection of saline to one side of the face
  Arms: control

SUMMARY:
This study is to evaluate the efficacy and tolerability of autologous adipose tissue derived stem cells in facial rejuvenation.

DETAILED DESCRIPTION:
Skin aging is a complex biological process that can be categorized into either extrinsic or intrinsic aging. Intrinsic aging is an inherent degenerative process caused by decreased proliferative capacity leading to cellular senescence. Extrinsic aging is caused by factors such as UV radiations, smoking and alcohol consumption.The physiological changes associated with aging of the skin are manifested in xerosis, dramatic loss of skin elasticity due to damage to collagen and elastin fibers; as well as barrier function, modification of rhytides and deficiencies in the regenerative property of the skin. All of which ultimately result in thinning of the skin, malar fat atrophy and pigmentary changes.Aging skin undergoes thinning of the epidermis that is caused by reduction of vascularity and hydration. On average, the thickness of the epidermis is reduced by about 6.4% during each decade of life.Skin aging effects can be assessed based on the skin appearance (texture and roughness, fine lines and wrinkles), structure, elasticity, hydration and barrier function. Many new non-invasive or minimally invasive bioengineering advances in recent years have enabled the quantitative analysis of skin properties during the aging processRecently, adult stem cells such as mesenchymal stem cells (MSCs) have been used in variable dermatologic conditions due to its regenerative properties such as wound healing, rejuvenation, acne scar and hair fall treatment. Different types of MSCs could be derived from different tissues as for example; bone marrow stem cells (BMSCs), adipose tissue-derived stem cells (ADSCs), and skin-derived stem cells (SDSCs)Adipose tissue derived stem cells are currently favorable compared to other types of adult stem cells as the procedure is easy, safe with minimal donor site morbidity. The process of obtaining a considerable amount of adipose tissues sufficient to use in skin regeneration is highly appealing due to its relative availability and accessibility. They secrete variable growth factors that affect surrounding environment as vascular endothelial growth factor (VEGF), platelet derived growth factor (PDGF), insulin like growth factors (IGF) and others

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed facial skin aging.
* Glogau photoaging score II and III.
* Body mass index ≥20 with adequate abdominal or other subcutaneous adipose tissue accessible for lipoaspiration.

Exclusion Criteria:

* History of keloid formation.
* Any coincidental chronic illness (e.g. metabolic, autoimmune or endocrinal) or malignancy.
* Any bleeding or coagulation disorder or recent use of anticoagulant therapy.
* Active infection.
* History of any previous aesthetic procedure on the face within the past 6 months.
* History of intake of anti-aging systemic or topical medications within the previous 3 months.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the degree of aesthetic improvement using the global aesthetic improvement scale GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse. | 6 months
  serial photography for assessment of degree of aesthetic improvement using the global aesthetic improvement scale GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse.

SECONDARY OUTCOMES:
Assessment of trans-epidermal water loss (TEWL) in gm /h-m2 using noninvasive probe (Dermal measurement system EDS12, UK) on both temple regions of the head | 6 months
  Assessment of trans-epidermal water loss (TEWL) in gm /h-m2 using noninvasive probe (Dermal measurement system EDS12, UK) on both temple regions of the head
Assessment of skin hydration in units using noninvasive probe (Dermal measurement system EDS12, UK) on both temple regions of the head | 6 months
  Assessment of hydration in units using noninvasive probe (Dermal measurement system EDS12, UK) on both temple regions of the head
Measurement of epidermal thickness in mm using UBM (Ultrasound Bio microscopy) on both temple regions of the head | 6 months
  Measurement of epidermal thickness in mm using UBM (Ultrasound Bio microscopy) on both temple regions of the head
Measurement of dermal thickness in mm using UBM (Ultrasound Bio microscopy) on both temple regions of the head | 6 months
  Measurement of dermal thickness in mm using UBM (Ultrasound Bio microscopy) on both temple regions of the head
A visual analog scale, will be used to assess participants' satisfaction by the treatment and side effects | 6 months
  A visual analog scale, will be used to assess participants' satisfaction by the treatment and side effects

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Ibrahim Farid Mohammed Amin, MD, Study Director — Assistant Professor of Dermatology, Faculty of Medicine, Alexandria University; Ossama Hussein Roshdy, MD, Study Director — Professor of Dermatology, Faculty of Medicine, Alexandria University; Wafaa Ibrahim Abdullah, MD, Study Director — Professor of Dermatology, Faculty of Medicine, Alexandria University; Radwa Ali Mehanna, PhD, Study Director — Assistant Professor of Physiology, Faculty of Medicine, Alexandria University; Nader Hussein Lotfy Bayoumi., MD, FRCS, Study Director — Professor of ophthalmology , Faculty of Medicine, Alexandria University
Locations (1):
- Aliaa Ismail, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03928444/Prot_000.pdf